CLINICAL TRIAL: NCT06479278
Title: Talk With Me Baby: Leveraging Well-Child Care to Enhance the Early Home Language Environment for Rural and Underserved Children
Brief Title: Talk With Me Baby to Enhance the Early Home Language Environment
Acronym: TWMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: National Institutes of Health (NIH) (NIH); University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 276453; U24OD024957 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Language Development; Speech; Infant Development; Infant Behavior; Language, Child; Language
MeSH Terms: conditions — Speech; Infant Behavior; Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Talk With Me Baby (Experimental)
  Interventions: Behavioral: Talk with Me Baby

INTERVENTIONS:
Behavioral: Talk with Me Baby — Primary care providers will embed Talk With Me Baby (TWMB) within standard-of-care Well-Child Care visits for children ≤36 months of age. Children will receive usual care plus a brief language-promotion intervention (TWMB) in up to 4 consecutive Well-Child Care visits during their 12-month period.

SUMMARY:
The goal of this clinical trial is to learn if the Talk With Me Baby (TWMB) program improves the home-language environment for at-risk families with children ages two to six months when primary care providers deliver the program during well-child checkups. The main question it aims to answer is:

Will the TWMB program increase the time a caregiver talks to their infant?

Participants will:

1. Come to at least four well-child checkups
2. Receive the TWMB program from the provider during the checkups
3. Record their conversations with their infant before they receive the program and after they receive the program four times.

ELIGIBILITY:
Inclusion Criteria:

For this study, each child-caregiver dyad will consist of:

1. A caregiver who will receive TWMB during routine WCC visits for their child at participating clinics, and
2. The child of the above caregiver for whom the WCC visits are conducted.

A potential caregiver participant must meet all the following inclusion criteria to enroll in the study:

1. Be the age of majority, or older, as defined by the state of residency.
2. Able to complete study measures in English.
3. Have the legal authority to consent to participate for themselves and to consent on behalf of their child.

To proceed to the follow-up portion of the study the caregiver (dyad) must have a LENA baseline assessment score that is ≤ 75th percentile compared to a child's age-referenced normative data.

A potential child participant must meet all the following inclusion criteria to be enrolled in the study:

1. Receive WCC at a participating clinic from a participating provider.
2. Be zero to nine months (+ 0-30 days) old at enrollment.
3. Was born at full term (> 37 weeks gestation).
4. Was born in a singleton birth (i.e., was the only child delivered during the birth).

Ages: 0 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in the home-language-environment promotion behaviors, as measured by the Language Environment Analysis (LENA) Conversational Turn Count percentile score from Baseline to Post-Intervention | 12 months
Improvement in the home-language-environment promotion behaviors, as measured by the Language Environment Analysis (LENA) Adult Word Count percentile score from Baseline to Post-Intervention | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kansas University Medical Center, Kansas City, Kansas
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Investigators will conduct this trial following the publication and data-sharing policies and regulations listed below:
  NIH Public Access Policy requires scientists to submit final peer-reviewed journal manuscripts arising from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  Environmental Influences on Child Health Outcomes (ECHO) IDeA States Pediatric Clinical Trials Network (ISPCTN) Publications and Presentations Policy ensures the accurate, responsible, and efficient communication of findings from ECHO ISPCTN clinical trials.
  NIH Data Sharing Policy and the policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Resulting Information Submission Rule. Other researchers may request data from this trial by contacting Song Ounpraseuth, Ph.D., at the ISPCTN Data Coordinating and Operations Center (DCOC).
Supporting Information: SAP, ICF
Time Frame: Per data sharing polices of NIH and the ISPCTN